CLINICAL TRIAL: NCT02451748
Title: IL-7 and IL-7R Expression in Peripheral Blood Mononuclear Cells, Peripheral Blood Monocytes or Differentiated Macrophages of Rheumatoid Arthritis Patients With Active vs. Inactive Disease Treated With DMARD and/or CIMZIA
Brief Title: IL-7 and IL-7R Expression in RA Patients With Active vs. Inactive Disease Treated With DMARD or CIMZIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Shiva Shahrara, Associate Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0117
Record Dates: First submitted 2015-05-06; First posted 2015-05-22 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Hydroxychloroquine; Sulfasalazine; Methylprednisolone; Prednisone; Triamcinolone; Naproxen; Leflunomide; Methotrexate; Adalimumab

STUDY DESIGN:
Intervention Model Description: In this study we determine whether expression of IL-7 and IL-7 receptor (R) is modulated by anti-tumor necrosis factor (TNF) treatment. For this purpose blood is obtained from RA patients prior to anti-TNF (Cimzia treatment; day 0) and after 3 months as well as 6 months of therapy. Transcription levels of IL-7 and IL-7R are examined from the peripheral blood obtained from day 0, 3 and 6 months of therapy. Results of this study will be reported in the MS in preparation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMARD's Responder and Non-Responder (Other): In the first group of subjects, blood samples will be obtained from (50) RA subjects with Disease modifying anti rheumatic drugs (DMARDs) such as methotrexate, plaquenil and/or prednisone that achieve remission (DAS28<2.6). The subjects that achieve remission (DAS28<2.6), blood will only be taken once at the subjects routine visit. Subject's that are non-responder to DMARDS will go onto group 2.
  Interventions: Other: Lab Work
- DMARD's plus Cimzia (Certolizumab pegol) (Other): The second group will consist of (150) RA subjects that did not respond to "DMARDs". These patients will further receive (DMARDs) such as methotrexate, plaquenil and/or prednisone as well as Cimzia®. In this Arm, blood samples will be collected onset of the study as well as 3 and 6 months after treatment with Cimzia at subject's visit through our collaboration with the aforementioned rheumatologists.
  Interventions: Other: Lab Work; Drug: Certolizumab pegol (CDP870, tradename Cimzia)(prefilled syringes at the dose of 200mg); Drug: Certolizumab pegol (CDP870, tradename Cimzia); Drug: Hydroxychloroquine; Drug: Sulfasalazine; Drug: Medrol; Drug: Prednisone; Drug: Triamcinolone; Drug: Naproxen; Drug: Leflunomide; Drug: Methotrexate; Drug: humira

INTERVENTIONS:
Other: Lab Work — Lab work to measure IL-7 and IL-7R
Drug: Certolizumab pegol (CDP870, tradename Cimzia)(prefilled syringes at the dose of 200mg) — Certolizumab pegol (CDP870, tradename Cimzia) or is provided in prefilled syringes at the dose of 200mg.
  Patients received 2x200mg at weeks 0, 2 and 4. Additionally a maintenance dose of 200mg is given every 2 weeks. Treatment is performed through subcutaneous injection.
  Other Names: Certolizumab pegol
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Certolizumab pegol (CDP870, tradename Cimzia) — rtolizumab pegol (CDP870, tradename Cimzia) or is provided in prefilled syringes at the dose of 200mg.
  Patients received 2x200mg at weeks 0, 2 and 4. Additionally a maintenance dose of 200mg is given every 2 weeks. Treatment is performed through subcutaneous injection.
  Other Names: Certolizumab pegol
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Hydroxychloroquine — some patients are on 400mg/day of hydroxychloroquine.
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Sulfasalazine — some patients are on 300 mg/day and some patients are on 1000 mg/day dose of sulfasalazine
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Medrol — some patients are on 8mg/day of medrol
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Prednisone — some patients are on 10mg /day, some patients are on 20 mg/day, some patients are on 2.5 mg/day, some patients are on 30 mg/day, and some patients are on 5 mg/day of prednisone
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Triamcinolone — some patients are on Triamcinolone 40-80mg IM monthly (received 40mg dose 1 week before blood draw, off enbrel 50mg weekly and SSZ 1000mg bid for ~ 3 months) some patients are on Triamcinolone 40mg IM monthly
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Naproxen — some patients are on 1000 mg/day of naproxen
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Leflunomide — some patients are on 20mg/day of leflunomide
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: Methotrexate — some patients are on 20mg weekly, some patients are on 25mg weekly, some patients are on 17.5 mg, some patients are on 15 mg weekly, some patients are on 7.5 mg weekly, and some patients are on 15 mg weekly dose of methotrexate
  Arms: DMARD's plus Cimzia (Certolizumab pegol)
Drug: humira — some patients are on Humira 40mg q2weeks
  Arms: DMARD's plus Cimzia (Certolizumab pegol)

SUMMARY:
The purpose of the study is to better understand the factors present in the cells of inflamed joints of patients with arthritis that may cause rheumatoid arthritis. Knowledge gained from this study may lead to new and better therapies for arthritis.

DETAILED DESCRIPTION:
Blood samples will be collected from patients that have been diagnosed with RA based on ACR classification criteria. The study will include 200 donors. The total number of subjects are divided into two groups to yield a power of 95% at a type I error 5% level [determined based on the preliminary data]. In the first group, 200 donors will be treated with methotrexate, plaquenil and/or prednisone (Disease modifying anti rheumatic drugs; DMARDs) that either achieve remission (Disease activity score, DAS28<2.6) or do not achieve remission (DAS28>2.6). 50 donor will be utilized as they respond to DMARDs and achieve remission (DAS28<2.6) and 150 donors that do not respond to DMARDs will be transferred to second group. In the second group, 150 donors will be treated with methotrexate, plaquenil and/or prednisone and Cimzia® (provided to us by UCB).

In the first group of patients, blood samples will be obtained from RA patients treated with Disease modifying anti rheumatic drugs (DMARDs) such as methotrexate, plaquenil and/or prednisone that achieve remission (DAS28<2.6). The patients that achieve remission (DAS28<2.6), blood will only be taken once at the patients routine visit.

The second group will consist of RA patients that did not respond to "DMARDs". These patients will further receive (DMARDs) such as methotrexate, plaquenil and/or prednisone as well as Cimzia® (provided to us by UCB) free of charge. Cimzia® is a FDA approved drug and is a standard of care. Blood samples will be obtained from the patients treated with DMARDs including methotrexate, plaquenil, and/or prednisone and Cimzia® (provided to us by UCB) that have inactive remission (DAS28<2.6). In this group, blood samples will be collected onset of the study as well as 3 and 6 months after treatment with Cimzia at patient's visit through our collaboration with the aforementioned rheumatologists. Patients receiving intra-articular steroid injections will be excluded from the study.

PB mononuclear cells will be isolated from RA whole blood and drawn into Blood collection tubes and isolated by Histopaque gradient centrifugation. Monocytes will be isolated from RA PB mononuclear cells by negative selection (as shown in the preliminary data) and half of the monocytes will be differentiated to macrophages for 7 days. The expression levels for IL-7 and IL-7R will be determined by real-time reverse transcription polymerase chain reaction (RT-PCR) and flow cytometry analysis.

In our statistical analysis, we will first perform a stratified analysis to evaluate the differential expression levels in RA patients with active and inactive disease, controlling for the type of treatment. Data analysis will be performed in collaboration with an UIC Center for Clinical and Translational Science statistician. Specifically, we will perform the comparison of IL-7 and IL-7R expression among RA patients with active (DAS28>2.6) vs. inactive disease (DAS28<2.6) for DMARDs group (group 1). We will then perform a similar comparison for the DMARDs and Cimzia® therapy group (group 2). The stratified analysis can adjust for the potential confounding effect of treatment received and allows for the detection of the potential differential relationships between expression levels of IL-7 or IL-7R and disease status. We will also perform a pooled regression analysis in which the expression logarithm of IL-7 or IL-7R from patients is regressed on the treatment group indicator [DMARDs (group 1) versus on DMARDs plus Cimzia® therapy (group 2)] and disease status (active or inactive disease) which would demonstrate the interaction between treatment groups and disease activity. Such an analysis pools subjects from two treatment groups together and can therefore increase the sample size, and hence potentially the power of detecting the relationships between biomarkers and disease status. The RA samples will be collected over a 2 year period and the data will be analyzed in the last year of the proposal.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet 1987 Revised Criteria for the Classification of Rheumatoid Arthritis defined as the diagnosis of the referring physician.
2. Persistent knee swelling (>ARA grade 2) for 2 weeks, and no recent intra-articular corticosteroid injection.
3. Age 18 years and older.
4. Must be on Disease modifying anti rheumatic drugs (DMARDs) such as methotrexate, plaquenil and/or prednisone.

Exclusion Criteria:

1. Patients having received intra-articular corticosteroid joint injection within the last 2-4 weeks.
2. Patients with active systemic or joint infections.
3. Women who are pregnant (pregnancy status will be self-reported)
4. Patients under 18 years of age
5. Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiva Shahrara, PhD, Principal Investigator — UIC
Locations (1):
- Outpatient Care Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Kim SJ, Chang HJ, Volin MV, Umar S, Van Raemdonck K, Chevalier A, Palasiewicz K, Christman JW, Volkov S, Arami S, Maz M, Mehta A, Zomorrodi RK, Fox DA, Sweiss N, Shahrara S. Macrophages are the primary effector cells in IL-7-induced arthritis. Cell Mol Immunol. 2020 Jul;17(7):728-740. doi: 10.1038/s41423-019-0235-z. Epub 2019 Jun 13. PMID 31197255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 10 patients were analyzed for IL-7 and IL-7R mRNA levels at onset, 3 months after Cimzia treatment and 6 months after Cimizia.
Groups:
- DMARD's Responder and Non-Responder: Individuals with rheumatoid arthritis (RA) receiving disease modifying anti-rheumatic drugs (DMARDs). Treating rheumatologists did not consistently measure DAS28<2.6, therefore this group consisted of both responders and non-responders to DMARDs (instead of only non-responders as originally planned). Blood samples were collected only once at the participant's routine visit.
- DMARD's Plus Cimzia (Certolizumab Pegol): Individuals with rheumatoid arthritis (RA) that did not respond to disease modifying anti-rheumatic drugs (DMARDs) were treated with DMARDs and Cimzia®. Cimzia® is an FDA approved drug and is a standard of care. In this group, blood samples were collected at study onset and 3 and 6 months after treatment with Cimzia at the patient's visit with the rheumatologists.
Period: Overall Study
Arm/Group | DMARD's Responder and Non-Responder | DMARD's Plus Cimzia (Certolizumab Pegol)
Started | 12 | 15
Participants With Evaluable Data at Visit 1 | 0 | 10
Participants With Evaluable Data at Visit 2 | 0 | 10
Participants With Evaluable Data at Visit 3 | 0 | 5
Completed | 0 | 5
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMARD's Responder and Non-Responder | DMARD's Plus Cimzia (Certolizumab Pegol) | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: IL-7 and IL-7R Expression in Peripheral Blood Mononuclear Cells of RA Patients With Active vs. Inactive Disease Treated With DMARD and/or CIMZIA.
Description: Expression of IL-7 and IL-7R mRNA levels measured by real-time RT-PCR.
Time Frame: baseline and 3 and 6 months
Population: 10 at 3 months, 5 at 6 months for DMARD's plus Cimzia group
Measure: Mean (Standard Error); unit: fold change vs housekeeping gene change
Groups:
- DMARD's Responder and Non-Responder: IL-7 and IL-7 receptor at baseline
- DMARD's Plus Cimzia (Certolizumab Pegol): IL-7 and IL-7 receptor at 3 and 6 months
Arm/Group | DMARD's Responder and Non-Responder | DMARD's Plus Cimzia (Certolizumab Pegol)
Number analyzed (Participants) | 0 | 10
fold change vs housekeeping gene change
  Visit 1 IL7 |  | 0.700 (0.132)
  Visit 1 IL7R |  | 1.330 (0.315)
  Visit 2 IL7 |  | 0.777 (0.104)
  Visit 2 IL7R |  | 1.460 (0.166)
  Visit 3 IL7: number analyzed (Participants) | 0 | 5
  Visit 3 IL7 |  | 0.569 (0.264)
  Visit 3 IL7R: number analyzed (Participants) | 0 | 5
  Visit 3 IL7R |  | 0.0163 (0.0157)
Statistical Analysis 1: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7 was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the first and second visit is as follows; Test type: Equivalence — ANOVA; p = 0.5378, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05
Statistical Analysis 2: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7 was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the first and third visit is as follows; Test type: Equivalence — ANOVA; p = 0.919, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05
Statistical Analysis 3: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7 was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the second and third visit is as follows; Test type: Equivalence — ANOVA; p = 0.4255, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05
Statistical Analysis 4: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7R was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the first and second visit is as follows; Test type: Equivalence — ANOVA; p = 0.1037, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05
Statistical Analysis 5: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7R was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the first and third visit is as follows; Test type: Equivalence — ANOVA; p = 0.0008, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05
Statistical Analysis 6: Comparison: DMARD's Plus Cimzia (Certolizumab Pegol); The mean mRNA expression for IL-7R was compared between all three visits simultaneously in RA Peripheral Blood Nonnuclear Cells. The comparison between the second and third visit is as follows; Test type: Equivalence — ANOVA; p = 0.0001, ANOVA — Tukey adjustment for multiple comparisons; A priori threshold was <0.05

ADVERSE EVENTS:
Time Frame: Adverse effects were assessed at 3 months (second visit) and 6 months (3rd visit).
Arm/Group | DMARD's Responder and Non-Responder | DMARD's Plus Cimzia (Certolizumab Pegol)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

LIMITATIONS AND CAVEATS:
Note - total participants = 10 -- same subjects proceeded from first arm to second arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02451748/Prot_SAP_000.pdf